CLINICAL TRIAL: NCT01156610
Title: Tobacco Treatment Outreach to Reduce Disparities for Primary Care Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer S. Haas, MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010P000405; P50CA148596 (NIH)
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Smoking; Smoking Cessation
Keywords: Smoking; Smoking Cessation; Electronic Health Record; Telephone
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Cessation Counseling (Experimental): IVR System: IVR will be used for two purposes: (1) to facilitate access to treatment for low-SES and minority smokers and (2) perform six-month outcome assessment.
  Tobacco Treatment Specialist Calls: A tobacco treatment specialist will make four attempts to contact the patient by phone within 14 days. On contacting the patient, the specialist will screen the patient for readiness to quit, provide brief (10 to 15 minutes) counseling tailored to the patient's readiness to quit, and provide information and support for use of medications that could be or were prescribed and about relevant community resources.
  NRT: Patients who do not have a contraindication and smoke > 10 cigarettes per day, will be offered a free 6-week kit of generic nicotine patches (2 weeks of 21 mg patches, 2 weeks of 14 mg patches, and 2 weeks of 7 mg patches). Individuals who smoke 5-10 cigarettes/day will be offered a 6-week course, starting with the 14 mg patch. Those with a contraindication will not get NRT.
  Interventions: Behavioral: Tobacco Treatment
- Usual Care (Active Comparator): IVR Call: Similar to the initial IVR call for the intervention arms, the initial control arm call will confirm the participant's identify and provide a brief description of the study (obtaining information about health behaviors), with the opportunity for the individual to accept or decline participation. Following this introduction, the IVR script will confirm smoking status. The phone script will collect specific information about current smoking (cigarettes/day), prior quit attempts, and motivation to quit during the next month. No further contact will be made with patients in the control clinics until the outcome assessment call. In the control practices, the IVR machine will also generate a text note documenting the information obtained for the patients' EHR for use by the patient's health care providers as part of their "visit-based" best practices.
  Interventions: Behavioral: Tobacco Treatment

INTERVENTIONS:
Behavioral: Tobacco Treatment — Comparison of integrated cessation counseling tools with the normal standard of care.
  Both the intervention and control clinics will be provided with tools for visit-based "best practices" for tobacco cessation. The LMR will provide smoking status icons and tobacco treatment reminders for the primary care physicians at the time of a visit. In addition, physicians in both arms have access to decision support around medications prescribed, including bupropion and varenicline. Physicians can refer patients to tobacco cessation groups that meet periodically at each of the sites or to the Massachusetts tobacco quitline.
  Outcome Assessment: Six month IVR Call: Patients in both the intervention and control practices who have not opted-out will be called six months after completing the 12-week treatment protocol. The outcome assessment script will be largely the same for intervention and control practices (except for the questions related to satisfaction with the intervention protocol).

SUMMARY:
The objectives of this project are to develop and evaluate a multi-level approach to tobacco treatment for low-SES and minority patients. The components of this intervention would include Integrated Voice Response(IVR)-facilitated systematic outreach, linkage to a tobacco treatment specialist, free Nicotine Replacement Therapy (NRT) directed at the patient, and integration of this program with both an individual's primary care physician through an electronic health record (EHR), as well as referral to community resources to address the socio-contextual barriers to tobacco cessation. To achieve these objectives, this intervention will test an innovative model of systematic outreach to low-SES and minority smokers using systematic phone outreach (including cell phones which are particularly prevalent among minority and low-SES groups), coordinated with the PCP, using both a cost-effective technology and a dedicated tobacco treatment specialist to increase smoking cessation in these populations. The proposed intervention will have multiple levels of influence (patient, PCP) and provide linkages to community resources. If successful, this model could be generalized to other health systems with an EHR, which are increasingly being promoted to improve the safety and quality of health care.

Hypothesis 1 (Reach and Effectiveness): An EHR-linked, IVR-mediated personalized treatment program for low-SES and minority smokers can reach these patients to increase quit rates and use of tobacco treatment effectively.

Hypothesis 2 (Adoption and Implementation): An EHR-linked, IVR-mediated personalized treatment program for low-SES and minority smokers can be adopted across a variety of practice settings and be consistently implemented across diverse patient populations.

DETAILED DESCRIPTION:
Because 70% of smokers have seen a PCP within the past year, primary care represents a valuable platform for reducing disparities in tobacco use that could be made more effective. The current national focus on expanding the use of EHRs also makes the proposed model to identify smokers with the goal of reducing disparities in tobacco use particularly timely. The adoption of EHRs in practices serving minorities is similar to that in all practices, suggesting that there is not a "digital divide" for PCP practices. In addition, the proposed intervention is novel because it addresses tobacco use at multiple levels (i.e., individual, health care setting, community), and is designed to provide smokers with tools to address socio-contextual contributors to disparities in tobacco use. Finally, the intervention will be informed by a broad approach using community resources for tobacco cessation. Conceptual models and empiric data suggest that this type of broad approach is needed to reach low-SES and minority smokers to reduce disparities in tobacco use. Telephone outreach may be particularly effective for minority and low-SES populations because cell phone penetration is higher in these populations. While disparities in tobacco use are rooted in social and economic problems that extend beyond the domain of health care and traditional treatment models, the health care system still represents a critical opportunity to initiate intervention.

Although smoking has declined over the past decades, substantial socioeconomic disparities in smoking prevalence, risk of addiction, and tobacco-related disease remain in the US, particularly among different racial, ethnic, and socioeconomic groups. Despite relatively similar rates of tobacco use, for example, African Americans (a term used interchangeably with "blacks" throughout this proposal) suffer from a higher burden of tobacco-related disease, particularly lung cancer, than whites. Importantly, low socioeconomic status (SES) and minority smokers also have a relatively more difficult time quitting for several reasons, including more limited access to treatment, misinformation about the risks and benefits of treatment, more environmental exposure, lack of social support, and other life stressors.

Primary care physicians (PCPs) are an important source of tobacco treatment, as the majority of smokers visit a PCP each year. While the US Public Health Service strongly recommends that clinicians identify and treat every tobacco user, such an approach is largely dependent on busy clinicians to provide counseling and treatment during a brief visit. Minority and low-SES smokers are more likely than whites to report that they did not receive counseling or treatment during a visit. For these reasons it is important to offer systematic opportunities for tobacco treatment beyond the provider's office, in addition to improving "best practices" for cessation treatment. Interactive Voice Response (IVR) is a phone technology that allows a computer to detect voice responses during a normal phone call (including calls from mobile phones). This technology offers a low-cost, efficient way to reach out proactively to large populations, independent of a visit. IVR scripts can be translated into other languages, facilitating systematic outreach to diverse populations. This technology can provide direct linkage to a tobacco treatment specialist, who can provide personalized advice for cessation, mood management, and stress reduction, and provide a course of free nicotine replacement treatment (NRT), as well as linkage to relevant community resources. Smokers who use NRT as part of their cessation plan are more likely to succeed than those who do not, and free NRT is a particularly important intervention for low-SES and minority smokers.

Specific Aim 1: To develop an EHR-linked, IVR-mediated personalized tobacco treatment program for low-SES and minority smokers. To develop this program, we will first conduct formative qualitative research to identify the particular barriers to smoking cessation faced by these populations and subsequently, to create a Community Resource Guide to address socio-cultural barriers to cessation.

Specific Aim 2: To measure the effectiveness of this personalized treatment program by conducting a randomized controlled trial of low-SES and minority smokers in 12 clinics from the Partners Primary Care Practice Based Research Network (PPC-PBRN). Patients in the intervention group will be offered three contacts with a tobacco treatment specialist over a 12 week period, a free 6-week supply of nicotine patches, and linkage to local resources using the Community Resource Guide. Patients in the control group will receive visit-based "best practices" care facilitated by EHR decision support (received by both the intervention and the control group). The primary outcome of this trial will be the 7-day abstinence rate at 6 months.

Specific Aim 3: To evaluate facilitators and barriers to the reach, adoption, and implementation of this personalized tobacco treatment program.

This project fits well with other projects in the Lung Cancer Disparities Center (LCDC), complementing the other projects that seek to explain disparities in lung cancer at the molecular, neighborhood, and societal levels. Over 80% of those diagnosed with lung cancer are current or ex-smokers, supporting the critical importance of smoking cessation to reducing disparities in lung cancer.1 Our project adds another layer by focusing on the individual/ clinical interface to reduce disparities in tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must be a current smoker.
* Must receive primary care at one of the participating clinics.
* Must have had a PCP visit within the last month at a participating clinic.
* Must have a working phone number listed in Partner's database.
* Must report race /ethnicity as African American or Hispanic or live in a low-SES block group (a census block group with a median income of < $65,000).
* Must speak English or Spanish.

Exclusion Criteria:

* Hearing impaired patients who cannot use the telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence of smoking six months following completion of the intervention protocol (nine months post randomization). | 2 years
  The difference between intervention and control patients ("smokers") who report nine months after randomization that they are now quitters (i.e., that they have not smoked for the past seven days but did smoke on enrollment). Self-reported smoking status has established validity when compared with measured serum cotinine levels and yields similar population prevalence estimates.

SECONDARY OUTCOMES:
Use of any Tobacco Treatment | 2 years
  The difference between intervention and control patients who report using any pharmacologic tobacco treatment (NRT replacement, bupropion, varenicline) or any behavioral treatment (state quitline, local tobacco program).
Use of Community Resources to Facilitate Smoking Cessation | 2 years
  The difference between intervention and control patients who report using community resources.
Patient Report of Socio-cultural Barriers to Tobacco Cessation | 2 years
  The difference between the percentage of intervention and control patients who report key socio-cultural barriers to tobacco cessation.
Quit Attempts | 2 years
  The difference between intervention and control patients who report making one or more quit attempts lasting >= 1 day during the nine months after randomization. An increasing number of quit attempts is related to ultimately quitting smoking. We will also examine difference in the number of quit attempts reported by the intervention and control groups within the nine months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Haas, MD, MSPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Molina JR, Yang P, Cassivi SD, Schild SE, Adjei AA. Non-small cell lung cancer: epidemiology, risk factors, treatment, and survivorship. Mayo Clin Proc. 2008 May;83(5):584-94. doi: 10.4065/83.5.584. PMID 18452692
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Background] Schroeder SA. Shattuck Lecture. We can do better--improving the health of the American people. N Engl J Med. 2007 Sep 20;357(12):1221-8. doi: 10.1056/NEJMsa073350. No abstract available. PMID 17881753
- [Background] Mendez D, Warner KE. Adult cigarette smoking prevalence: declining as expected (not as desired). Am J Public Health. 2004 Feb;94(2):251-2. doi: 10.2105/ajph.94.2.251. PMID 14759934
- [Background] Rigotti NA. Clinical practice. Treatment of tobacco use and dependence. N Engl J Med. 2002 Feb 14;346(7):506-12. doi: 10.1056/NEJMcp012279. No abstract available. PMID 11844853
- [Background] Meara ER, Richards S, Cutler DM. The gap gets bigger: changes in mortality and life expectancy, by education, 1981-2000. Health Aff (Millwood). 2008 Mar-Apr;27(2):350-60. doi: 10.1377/hlthaff.27.2.350. PMID 18332489
- [Background] Haiman CA, Stram DO, Wilkens LR, Pike MC, Kolonel LN, Henderson BE, Le Marchand L. Ethnic and racial differences in the smoking-related risk of lung cancer. N Engl J Med. 2006 Jan 26;354(4):333-42. doi: 10.1056/NEJMoa033250. PMID 16436765
- [Background] Harman J, Graham H, Francis B, Inskip HM; SWS Study Group. Socioeconomic gradients in smoking among young women: A British survey. Soc Sci Med. 2006 Dec;63(11):2791-800. doi: 10.1016/j.socscimed.2006.07.021. Epub 2006 Sep 7. PMID 16962221
- [Background] Gruer L, Hart CL, Gordon DS, Watt GC. Effect of tobacco smoking on survival of men and women by social position: a 28 year cohort study. BMJ. 2009 Feb 17;338:b480. doi: 10.1136/bmj.b480. PMID 19224884
- [Background] Murphy JM, Mahoney MC, Hyland AJ, Higbee C, Cummings KM. Disparity in the use of smoking cessation pharmacotherapy among Medicaid and general population smokers. J Public Health Manag Pract. 2005 Jul-Aug;11(4):341-5. doi: 10.1097/00124784-200507000-00013. PMID 15958934
- [Background] Honjo K, Tsutsumi A, Kawachi I, Kawakami N. What accounts for the relationship between social class and smoking cessation? Results of a path analysis. Soc Sci Med. 2006 Jan;62(2):317-28. doi: 10.1016/j.socscimed.2005.06.011. Epub 2005 Jul 21. PMID 16039765
- [Background] Jaen CR, Cummings KM, Shah D, Aungst W. Patterns of use of a free nicotine patch program for Medicaid and uninsured patients. J Natl Med Assoc. 1997 May;89(5):325-8. PMID 9170833
- [Background] Cummings KM, Hyland A, Giovino GA, Hastrup JL, Bauer JE, Bansal MA. Are smokers adequately informed about the health risks of smoking and medicinal nicotine? Nicotine Tob Res. 2004 Dec;6 Suppl 3:S333-40. doi: 10.1080/14622200412331320734. PMID 15799596
- [Background] Lee D, Turner N, Burns J, Lee T. Tobacco use and low-income African Americans: policy implications. Addict Behav. 2007 Feb;32(2):332-41. doi: 10.1016/j.addbeh.2006.05.002. Epub 2006 Jul 7. PMID 16828978
- [Background] Graham AL, Papandonatos GD, DePue JD, Pinto BM, Borrelli B, Neighbors CJ, Niaura R, Buka SL, Abrams DB. Lifetime characteristics of participants and non-participants in a smoking cessation trial: implications for external validity and public health impact. Ann Behav Med. 2008 Jun;35(3):295-307. doi: 10.1007/s12160-008-9031-1. Epub 2008 Apr 15. PMID 18414962
- [Background] Manfredi C, Lacey LP, Warnecke R, Petraitis J. Sociopsychological correlates of motivation to quit smoking among low-SES African American women. Health Educ Behav. 1998 Jun;25(3):304-18. doi: 10.1177/109019819802500306. PMID 9615241
- [Background] Lacey LP, Manfredi C, Balch G, Warnecke RB, Allen K, Edwards C. Social support in smoking cessation among black women in Chicago public housing. Public Health Rep. 1993 May-Jun;108(3):387-94. PMID 8497578
- [Background] Stead M, MacAskill S, MacKintosh AM, Reece J, Eadie D. "It's as if you're locked in": qualitative explanations for area effects on smoking in disadvantaged communities. Health Place. 2001 Dec;7(4):333-43. doi: 10.1016/s1353-8292(01)00025-9. PMID 11682332
- [Background] Barbeau EM, Wolin KY, Naumova EN, Balbach E. Tobacco advertising in communities: associations with race and class. Prev Med. 2005 Jan;40(1):16-22. doi: 10.1016/j.ypmed.2004.04.056. PMID 15530576
- [Background] Lynch JW, Kaplan GA, Salonen JT. Why do poor people behave poorly? Variation in adult health behaviours and psychosocial characteristics by stages of the socioeconomic lifecourse. Soc Sci Med. 1997 Mar;44(6):809-19. doi: 10.1016/s0277-9536(96)00191-8. PMID 9080564
- [Background] Webb MS, Carey MP. Tobacco smoking among low-income Black women: demographic and psychosocial correlates in a community sample. Nicotine Tob Res. 2008 Jan;10(1):219-29. doi: 10.1080/14622200701767845. PMID 18188763
- [Background] Barbeau EM, Krieger N, Soobader MJ. Working class matters: socioeconomic disadvantage, race/ethnicity, gender, and smoking in NHIS 2000. Am J Public Health. 2004 Feb;94(2):269-78. doi: 10.2105/ajph.94.2.269. PMID 14759942
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette use among high school students--United States, 1991-2007. MMWR Morb Mortal Wkly Rep. 2008 Jun 27;57(25):686-8. PMID 18583955
- [Background] Perez-Stable EJ, Herrera B, Jacob P 3rd, Benowitz NL. Nicotine metabolism and intake in black and white smokers. JAMA. 1998 Jul 8;280(2):152-6. doi: 10.1001/jama.280.2.152. PMID 9669788
- [Background] Benowitz NL. Clinical pharmacology of nicotine: implications for understanding, preventing, and treating tobacco addiction. Clin Pharmacol Ther. 2008 Apr;83(4):531-41. doi: 10.1038/clpt.2008.3. Epub 2008 Feb 27. PMID 18305452
- [Background] Kreslake JM, Wayne GF, Connolly GN. The menthol smoker: tobacco industry research on consumer sensory perception of menthol cigarettes and its role in smoking behavior. Nicotine Tob Res. 2008 Apr;10(4):705-15. doi: 10.1080/14622200801979134. PMID 18418792
- [Background] Pletcher MJ, Hulley BJ, Houston T, Kiefe CI, Benowitz N, Sidney S. Menthol cigarettes, smoking cessation, atherosclerosis, and pulmonary function: the Coronary Artery Risk Development in Young Adults (CARDIA) Study. Arch Intern Med. 2006 Sep 25;166(17):1915-22. doi: 10.1001/archinte.166.17.1915. PMID 17000950
- [Background] Gandhi KK, Foulds J, Steinberg MB, Lu SE, Williams JM. Lower quit rates among African American and Latino menthol cigarette smokers at a tobacco treatment clinic. Int J Clin Pract. 2009 Mar;63(3):360-7. doi: 10.1111/j.1742-1241.2008.01969.x. PMID 19222622
- [Background] Bennett GG, Wolin KY, Robinson EL, Fowler S, Edwards CL. Perceived racial/ethnic harassment and tobacco use among African American young adults. Am J Public Health. 2005 Feb;95(2):238-40. doi: 10.2105/AJPH.2004.037812. PMID 15671457
- [Background] Lopez-Quintero C, Crum RM, Neumark YD. Racial/ethnic disparities in report of physician-provided smoking cessation advice: analysis of the 2000 National Health Interview Survey. Am J Public Health. 2006 Dec;96(12):2235-9. doi: 10.2105/AJPH.2005.071035. Epub 2006 Jun 29. PMID 16809587
- [Background] Cokkinides VE, Halpern MT, Barbeau EM, Ward E, Thun MJ. Racial and ethnic disparities in smoking-cessation interventions: analysis of the 2005 National Health Interview Survey. Am J Prev Med. 2008 May;34(5):404-12. doi: 10.1016/j.amepre.2008.02.003. PMID 18407007
- [Background] Sonnenfeld N, Schappert SM, Lin SX. Racial and ethnic differences in delivery of tobacco-cessation services. Am J Prev Med. 2009 Jan;36(1):21-8. doi: 10.1016/j.amepre.2008.09.028. Epub 2008 Nov 1. PMID 18977111
- [Background] Wong MD, Ettner SL, Boscardin WJ, Shapiro MF. The contribution of cancer incidence, stage at diagnosis and survival to racial differences in years of life expectancy. J Gen Intern Med. 2009 Apr;24(4):475-81. doi: 10.1007/s11606-009-0912-1. Epub 2009 Feb 3. PMID 19189193
- [Background] Wilson K, Gibson N, Willan A, Cook D. Effect of smoking cessation on mortality after myocardial infarction: meta-analysis of cohort studies. Arch Intern Med. 2000 Apr 10;160(7):939-44. doi: 10.1001/archinte.160.7.939. PMID 10761958
- [Background] LaCroix AZ, Lang J, Scherr P, Wallace RB, Cornoni-Huntley J, Berkman L, Curb JD, Evans D, Hennekens CH. Smoking and mortality among older men and women in three communities. N Engl J Med. 1991 Jun 6;324(23):1619-25. doi: 10.1056/NEJM199106063242303. PMID 2030718
- [Background] Tsevat J. Impact and cost-effectiveness of smoking interventions. Am J Med. 1992 Jul 15;93(1A):43S-47S. doi: 10.1016/0002-9343(92)90627-n. PMID 1497003
- [Background] Anthonisen NR, Skeans MA, Wise RA, Manfreda J, Kanner RE, Connett JE; Lung Health Study Research Group. The effects of a smoking cessation intervention on 14.5-year mortality: a randomized clinical trial. Ann Intern Med. 2005 Feb 15;142(4):233-9. doi: 10.7326/0003-4819-142-4-200502150-00005. PMID 15710956
- [Background] Cromwell J, Bartosch WJ, Fiore MC, Hasselblad V, Baker T. Cost-effectiveness of the clinical practice recommendations in the AHCPR guideline for smoking cessation. Agency for Health Care Policy and Research. JAMA. 1997 Dec 3;278(21):1759-66. PMID 9388153
- [Background] Westmaas JL, Langsam K. Unaided smoking cessation and predictors of failure to quit in a community sample: effects of gender. Addict Behav. 2005 Aug;30(7):1405-24. doi: 10.1016/j.addbeh.2005.03.001. PMID 15896921
- [Background] Cahill K, Stead LF, Lancaster T. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD006103. doi: 10.1002/14651858.CD006103.pub2. PMID 17253581
- [Background] Cokkinides VE, Ward E, Jemal A, Thun MJ. Under-use of smoking-cessation treatments: results from the National Health Interview Survey, 2000. Am J Prev Med. 2005 Jan;28(1):119-22. doi: 10.1016/j.amepre.2004.09.007. PMID 15626567
- [Background] Browning KK, Ferketich AK, Salsberry PJ, Wewers ME. Socioeconomic disparity in provider-delivered assistance to quit smoking. Nicotine Tob Res. 2008 Jan;10(1):55-61. doi: 10.1080/14622200701704905. PMID 18188745
- [Background] Shiffman S, Brockwell SE, Pillitteri JL, Gitchell JG. Use of smoking-cessation treatments in the United States. Am J Prev Med. 2008 Feb;34(2):102-11. doi: 10.1016/j.amepre.2007.09.033. PMID 18201639
- [Background] Orleans CT. Increasing the demand for and use of effective smoking-cessation treatments reaping the full health benefits of tobacco-control science and policy gains--in our lifetime. Am J Prev Med. 2007 Dec;33(6 Suppl):S340-8. doi: 10.1016/j.amepre.2007.09.003. PMID 18021909
- [Background] Fu SS, Kodl MM, Joseph AM, Hatsukami DK, Johnson EO, Breslau N, Wu B, Bierut L. Racial/Ethnic disparities in the use of nicotine replacement therapy and quit ratios in lifetime smokers ages 25 to 44 years. Cancer Epidemiol Biomarkers Prev. 2008 Jul;17(7):1640-7. doi: 10.1158/1055-9965.EPI-07-2726. Epub 2008 Jun 26. PMID 18583471
- [Background] Fu SS, Sherman SE, Yano EM, van Ryn M, Lanto AB, Joseph AM. Ethnic disparities in the use of nicotine replacement therapy for smoking cessation in an equal access health care system. Am J Health Promot. 2005 Nov-Dec;20(2):108-16. doi: 10.4278/0890-1171-20.2.108. PMID 16295702
- [Background] Fu SS, Burgess D, van Ryn M, Hatsukami DK, Solomon J, Joseph AM. Views on smoking cessation methods in ethnic minority communities: a qualitative investigation. Prev Med. 2007 Mar;44(3):235-40. doi: 10.1016/j.ypmed.2006.11.002. Epub 2006 Dec 18. PMID 17175016
- [Background] Yerger VB, Przewoznik J, Malone RE. Racialized geography, corporate activity, and health disparities: tobacco industry targeting of inner cities. J Health Care Poor Underserved. 2007 Nov;18(4 Suppl):10-38. doi: 10.1353/hpu.2007.0120. PMID 18065850
- [Background] Vardavas CI, Connolly GN, Kafatos AG. Geographical information systems as a tool for monitoring tobacco industry advertising. Tob Control. 2009 Jun;18(3):190-6. doi: 10.1136/tc.2008.026856. Epub 2009 Feb 2. PMID 19188209
- [Background] Primack BA, Bost JE, Land SR, Fine MJ. Volume of tobacco advertising in African American markets: systematic review and meta-analysis. Public Health Rep. 2007 Sep-Oct;122(5):607-15. doi: 10.1177/003335490712200508. PMID 17877308
- [Background] Wiltshire S, Bancroft A, Parry O, Amos A. 'I came back here and started smoking again': perceptions and experiences of quitting among disadvantaged smokers. Health Educ Res. 2003 Jun;18(3):292-303. doi: 10.1093/her/cyf031. PMID 12828231
- [Background] Stead LF, Lancaster T. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2001;(2):CD002850. doi: 10.1002/14651858.CD002850. PMID 11406050
- [Background] Lawrence D, Graber JE, Mills SL, Meissner HI, Warnecke R. Smoking cessation interventions in U.S. racial/ethnic minority populations: an assessment of the literature. Prev Med. 2003 Feb;36(2):204-16. doi: 10.1016/s0091-7435(02)00023-3. PMID 12590996
- [Background] Miller CL, Sedivy V. Using a quitline plus low-cost nicotine replacement therapy to help disadvantaged smokers to quit. Tob Control. 2009 Apr;18(2):144-9. doi: 10.1136/tc.2008.026492. Epub 2009 Jan 8. PMID 19131454
- [Background] Maher JE, Rohde K, Dent CW, Stark MJ, Pizacani B, Boysun MJ, Dilley JA, Yepassis-Zembrou PL. Is a statewide tobacco quitline an appropriate service for specific populations? Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i65-70. doi: 10.1136/tc.2006.019786. PMID 18048635
- [Background] Fernander AF, Patten CA, Schroeder DR, Stevens SR, Croghan IT, Offord KP, Hurt RD. Characteristics of six-month tobacco use outcomes of Black patients seeking smoking cessation intervention. J Health Care Poor Underserved. 2006 May;17(2):413-24. doi: 10.1353/hpu.2006.0059. PMID 16702724
- [Background] Ockene JK, Kristeller J, Goldberg R, Amick TL, Pekow PS, Hosmer D, Quirk M, Kalan K. Increasing the efficacy of physician-delivered smoking interventions: a randomized clinical trial. J Gen Intern Med. 1991 Jan-Feb;6(1):1-8. doi: 10.1007/BF02599381. PMID 1999742
- [Background] Thorndike AN, Regan S, Rigotti NA. The treatment of smoking by US physicians during ambulatory visits: 1994 2003. Am J Public Health. 2007 Oct;97(10):1878-83. doi: 10.2105/AJPH.2006.092577. Epub 2007 Aug 29. PMID 17761570
- [Background] Schroeder SA. What to do with a patient who smokes. JAMA. 2005 Jul 27;294(4):482-7. doi: 10.1001/jama.294.4.482. PMID 16046655
- [Background] Hollis JF, Bills R, Whitlock E, Stevens VJ, Mullooly J, Lichtenstein E. Implementing tobacco interventions in the real world of managed care. Tob Control. 2000;9 Suppl 1(Suppl 1):I18-24. doi: 10.1136/tc.9.suppl_1.i18. No abstract available. PMID 10688926
- [Background] Lichtenstein E, Hollis JF, Severson HH, Stevens VJ, Vogt TM, Glasgow RE, Andrews JA. Tobacco cessation interventions in health care settings: rationale, model, outcomes. Addict Behav. 1996 Nov-Dec;21(6):709-20. doi: 10.1016/0306-4603(96)00030-5. PMID 8904937
- [Background] Frieden TR, Mostashari F, Kerker BD, Miller N, Hajat A, Frankel M. Adult tobacco use levels after intensive tobacco control measures: New York City, 2002-2003. Am J Public Health. 2005 Jun;95(6):1016-23. doi: 10.2105/AJPH.2004.058164. PMID 15914827
- [Background] McDaniel AM, Benson PL, Roesener GH, Martindale J. An integrated computer-based system to support nicotine dependence treatment in primary care. Nicotine Tob Res. 2005 Apr;7 Suppl 1:S57-66. doi: 10.1080/14622200500078139. PMID 16036271
- [Background] Forster AJ, LaBranche R, McKim R, Faught JW, Feasby TE, Janes-Kelley S, Shojania KG, van Walraven C. Automated patient assessments after outpatient surgery using an interactive voice response system. Am J Manag Care. 2008 Jul;14(7):429-36. PMID 18611094
- [Background] Piette JD, Weinberger M, Kraemer FB, McPhee SJ. Impact of automated calls with nurse follow-up on diabetes treatment outcomes in a Department of Veterans Affairs Health Care System: a randomized controlled trial. Diabetes Care. 2001 Feb;24(2):202-8. doi: 10.2337/diacare.24.2.202. PMID 11213866
- [Background] Piette JD, Weinberger M, McPhee SJ. The effect of automated calls with telephone nurse follow-up on patient-centered outcomes of diabetes care: a randomized, controlled trial. Med Care. 2000 Feb;38(2):218-30. doi: 10.1097/00005650-200002000-00011. PMID 10659695
- [Background] Farzanfar R, Finkelstein J, Friedman RH. Testing the usability of two automated home-based patient-management systems. J Med Syst. 2004 Apr;28(2):143-53. doi: 10.1023/b:joms.0000023297.50379.3c. PMID 15195845
- [Background] Friedman RH, Kazis LE, Jette A, Smith MB, Stollerman J, Torgerson J, Carey K. A telecommunications system for monitoring and counseling patients with hypertension. Impact on medication adherence and blood pressure control. Am J Hypertens. 1996 Apr;9(4 Pt 1):285-92. doi: 10.1016/0895-7061(95)00353-3. PMID 8722429
- [Background] Adams WG, Wright JA, Noland CM, Watson BL, Friedman RH. TLC-HEAT: Telephony-based self-care for overweight children. AMIA Annu Symp Proc. 2007 Oct 11:859. PMID 18693961
- [Background] Migneault JP, Farzanfar R, Wright JA, Friedman RH. How to write health dialog for a talking computer. J Biomed Inform. 2006 Oct;39(5):468-81. doi: 10.1016/j.jbi.2006.02.009. Epub 2006 Feb 23. PMID 16564749
- [Background] Friedman RH. Automated telephone conversations to assess health behavior and deliver behavioral interventions. J Med Syst. 1998 Apr;22(2):95-102. doi: 10.1023/a:1022695119046. PMID 9571516
- [Background] Friedman RH, Stollerman J, Rozenblyum L, Belfer D, Selim A, Mahoney D, Steinbach S. A telecommunications system to manage patients with chronic disease. Stud Health Technol Inform. 1998;52 Pt 2:1330-4. PMID 10384677
- [Background] Toll BA, Cooney NL, McKee SA, O'Malley SS. Correspondence between Interactive Voice Response (IVR) and Timeline Followback (TLFB) reports of drinking behavior. Addict Behav. 2006 Apr;31(4):726-31. doi: 10.1016/j.addbeh.2005.05.044. Epub 2005 Jun 21. PMID 15975732
- [Background] Piette JD, McPhee SJ, Weinberger M, Mah CA, Kraemer FB. Use of automated telephone disease management calls in an ethnically diverse sample of low-income patients with diabetes. Diabetes Care. 1999 Aug;22(8):1302-9. doi: 10.2337/diacare.22.8.1302. PMID 10480775
- [Background] Goldman RE, Sanchez-Hernandez M, Ross-Degnan D, Piette JD, Trinacty CM, Simon SR. Developing an automated speech-recognition telephone diabetes intervention. Int J Qual Health Care. 2008 Aug;20(4):264-70. doi: 10.1093/intqhc/mzn021. Epub 2008 May 20. PMID 18492706
- [Background] Killen JD, Fortmann SP, Schatzberg AF, Hayward C, Sussman L, Rothman M, Strausberg L, Varady A. Nicotine patch and paroxetine for smoking cessation. J Consult Clin Psychol. 2000 Oct;68(5):883-9. PMID 11068974
- [Background] Shiffman S, Dresler CM, Hajek P, Gilburt SJ, Targett DA, Strahs KR. Efficacy of a nicotine lozenge for smoking cessation. Arch Intern Med. 2002 Jun 10;162(11):1267-76. doi: 10.1001/archinte.162.11.1267. PMID 12038945
- [Background] Brendryen H, Drozd F, Kraft P. A digital smoking cessation program delivered through internet and cell phone without nicotine replacement (happy ending): randomized controlled trial. J Med Internet Res. 2008 Nov 28;10(5):e51. doi: 10.2196/jmir.1005. PMID 19087949
- [Background] Brendryen H, Kraft P. Happy ending: a randomized controlled trial of a digital multi-media smoking cessation intervention. Addiction. 2008 Mar;103(3):478-84; discussion 485-6. doi: 10.1111/j.1360-0443.2007.02119.x. PMID 18269367
- [Background] Regan S, Reyen M, Lockhart AC, Richards AE, Rigotti NA. Using Interactive Voice Recognition Technology to Assess Smoking Outcomes and Link Smokers to Counseling after Hospital Discharge. Paper presented at: 2009 Annual Meeting, Society for Research in Nicotine and Tobacco, 2009; Dublin, Ireland.
- [Background] Wagner EH, Austin BT, Von Korff M. Improving outcomes in chronic illness. Manag Care Q. 1996 Spring;4(2):12-25. PMID 10157259
- [Background] Wagner EH, Austin BT, Von Korff M. Organizing care for patients with chronic illness. Milbank Q. 1996;74(4):511-44. PMID 8941260
- [Background] Katz ML, Sheridan S, Pignone M, Lewis C, Battle J, Gollop C, O'Malley M. Prostate and colon cancer screening messages in popular magazines. J Gen Intern Med. 2004 Aug;19(8):843-8. doi: 10.1111/j.1525-1497.2004.30504.x. PMID 15242469
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Glasgow RE, Bull SS, Gillette C, Klesges LM, Dzewaltowski DA. Behavior change intervention research in healthcare settings: a review of recent reports with emphasis on external validity. Am J Prev Med. 2002 Jul;23(1):62-9. doi: 10.1016/s0749-3797(02)00437-3. PMID 12093425
- [Background] Dzewaltowski DA, Glasgow RE, Klesges LM, Estabrooks PA, Brock E. RE-AIM: evidence-based standards and a Web resource to improve translation of research into practice. Ann Behav Med. 2004 Oct;28(2):75-80. doi: 10.1207/s15324796abm2802_1. PMID 15454353
- [Background] Eakin EG, Brown WJ, Marshall AL, Mummery K, Larsen E. Physical activity promotion in primary care: bridging the gap between research and practice. Am J Prev Med. 2004 Nov;27(4):297-303. doi: 10.1016/j.amepre.2004.07.012. PMID 15488359
- [Background] Sorensen G, Barbeau E, Hunt MK, Emmons K. Reducing social disparities in tobacco use: a social-contextual model for reducing tobacco use among blue-collar workers. Am J Public Health. 2004 Feb;94(2):230-9. doi: 10.2105/ajph.94.2.230. PMID 14759932
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Ajzen I, Fishbein M. Understanding attitudes and predicting social behavior. Englewood Cliffs, N.J.: Prentice Hall; 1980.
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Jha AK, Bates DW, Jenter C, Orav EJ, Zheng J, Cleary P, Simon SR. Electronic health records: use, barriers and satisfaction among physicians who care for black and Hispanic patients. J Eval Clin Pract. 2009 Feb;15(1):158-63. doi: 10.1111/j.1365-2753.2008.00975.x. Epub 2008 Aug 28. PMID 18759752
- [Background] Williams DR, Collins C. US socioeconomic and racial differences in health: patterns and explanations. Annual Review of Sociology. Vol 21; 1995:349 (338 pages).
- [Background] Williams DR. Race, socioeconomic status, and health. The added effects of racism and discrimination. Ann N Y Acad Sci. 1999;896:173-88. doi: 10.1111/j.1749-6632.1999.tb08114.x. PMID 10681897
- [Background] Williams DR, Rucker TD. Understanding and addressing racial disparities in health care. Health Care Financ Rev. 2000 Summer;21(4):75-90. PMID 11481746
- [Background] Williams DR, Lavizzo-Mourey R, Warren RC. The concept of race and health status in America. Public Health Rep. 1994 Jan-Feb;109(1):26-41. PMID 8303011
- [Background] Williams DR, Jackson PB. Social sources of racial disparities in health. Health Aff (Millwood). 2005 Mar-Apr;24(2):325-34. doi: 10.1377/hlthaff.24.2.325. PMID 15757915
- [Background] Williams DR, Jackson JS. Race/ethnicity and the 2000 census: recommendations for African American and other black populations in the United States. Am J Public Health. 2000 Nov;90(11):1728-30. doi: 10.2105/ajph.90.11.1728. PMID 11076240
- [Background] Williams DR, Haile R, Gonzalez HM, Neighbors H, Baser R, Jackson JS. The mental health of Black Caribbean immigrants: results from the National Survey of American Life. Am J Public Health. 2007 Jan;97(1):52-9. doi: 10.2105/AJPH.2006.088211. Epub 2006 Nov 30. PMID 17138909
- [Background] Williams DR, Collins C. Racial residential segregation: a fundamental cause of racial disparities in health. Public Health Rep. 2001 Sep-Oct;116(5):404-16. doi: 10.1093/phr/116.5.404. PMID 12042604
- [Background] Williams DR. The health of U.S. racial and ethnic populations. J Gerontol B Psychol Sci Soc Sci. 2005 Oct;60 Spec No 2:53-62. doi: 10.1093/geronb/60.special_issue_2.s53. PMID 16251591
- [Background] De Jesus M. Mutuality at the center: health promotion with Cape Verdean immigrant women. Ethn Health. 2009 Feb;14(1):45-59. doi: 10.1080/13557850802023141. PMID 19152158
- [Background] De Jesus M. The importance of social context in understanding and promoting low-income immigrant women's health. J Health Care Poor Underserved. 2009 Feb;20(1):90-7. doi: 10.1353/hpu.0.0126. PMID 19202249
- [Background] De Jesus M. Institutional barriers and strategies to health promotion: perspectives and experiences of Cape Verdean women health promoters. J Immigr Minor Health. 2010 Jun;12(3):398-407. doi: 10.1007/s10903-008-9127-5. Epub 2008 Feb 29. PMID 18307042
- [Background] McWilliams JM, Meara E, Zaslavsky AM, Ayanian JZ. Differences in control of cardiovascular disease and diabetes by race, ethnicity, and education: U.S. trends from 1999 to 2006 and effects of medicare coverage. Ann Intern Med. 2009 Apr 21;150(8):505-15. doi: 10.7326/0003-4819-150-8-200904210-00005. PMID 19380852
- [Background] Kang-Kim M, Betancourt JR, Ayanian JZ, Zaslavsky AM, Yucel RM, Weissman JS. Access to care and use of preventive services by Hispanics: state-based variations from 1991 to 2004. Med Care. 2008 May;46(5):507-15. doi: 10.1097/MLR.0b013e31816dd966. PMID 18438199
- [Background] McGuire TG, Ayanian JZ, Ford DE, Henke RE, Rost KM, Zaslavsky AM. Testing for statistical discrimination by race/ethnicity in panel data for depression treatment in primary care. Health Serv Res. 2008 Apr;43(2):531-51. doi: 10.1111/j.1475-6773.2007.00770.x. PMID 18370966
- [Background] Gilman SE, Breslau J, Conron KJ, Koenen KC, Subramanian SV, Zaslavsky AM. Education and race-ethnicity differences in the lifetime risk of alcohol dependence. J Epidemiol Community Health. 2008 Mar;62(3):224-30. doi: 10.1136/jech.2006.059022. PMID 18272737
- [Background] Trivedi AN, Zaslavsky AM, Schneider EC, Ayanian JZ. Relationship between quality of care and racial disparities in Medicare health plans. JAMA. 2006 Oct 25;296(16):1998-2004. doi: 10.1001/jama.296.16.1998. PMID 17062863
- [Background] Keating NL, Herrinton LJ, Zaslavsky AM, Liu L, Ayanian JZ. Variations in hospice use among cancer patients. J Natl Cancer Inst. 2006 Aug 2;98(15):1053-9. doi: 10.1093/jnci/djj298. PMID 16882942
- [Background] Trivedi AN, Zaslavsky AM, Schneider EC, Ayanian JZ. Trends in the quality of care and racial disparities in Medicare managed care. N Engl J Med. 2005 Aug 18;353(7):692-700. doi: 10.1056/NEJMsa051207. PMID 16107622
- [Background] Schneider EC, Zaslavsky AM, Epstein AM. Racial disparities in the quality of care for enrollees in medicare managed care. JAMA. 2002 Mar 13;287(10):1288-94. doi: 10.1001/jama.287.10.1288. PMID 11886320
- [Background] Geller AC, Lash TL, Siegel B, Annas GD, Prout MN. The primary care pediatrician's influence on medical student's performance of smoking assessments and counseling. Prev Med. 2005 Jul;41(1):47-52. doi: 10.1016/j.ypmed.2004.08.002. Epub 2004 Nov 10. PMID 15916992
- [Background] Winickoff JP, Berkowitz AB, Brooks K, Tanski SE, Geller A, Thomson C, Lando HA, Curry S, Muramoto M, Prokhorov AV, Best D, Weitzman M, Pbert L; Tobacco Consortium, Center for Child Health Research of the American Academy of Pediatrics. State-of-the-art interventions for office-based parental tobacco control. Pediatrics. 2005 Mar;115(3):750-60. doi: 10.1542/peds.2004-1055. PMID 15741382
- [Background] Geller AC, Emmons KM, Brooks DR, Powers C, Zhang Z, Koh HK, Heeren T, Sober AJ, Li F, Gilchrest BA. A randomized trial to improve early detection and prevention practices among siblings of melanoma patients. Cancer. 2006 Aug 15;107(4):806-14. doi: 10.1002/cncr.22050. PMID 16832795
- [Background] Geller AC, Brooks DR, Powers CA, Brooks KR, Rigotti NA, Bognar B, McIntosh S, Zapka J. Tobacco cessation and prevention practices reported by second and fourth year students at US medical schools. J Gen Intern Med. 2008 Jul;23(7):1071-6. doi: 10.1007/s11606-008-0526-z. PMID 18612747
- [Background] Powers CA, Thomson CC, Feuerstein I, Cross M, Powers EM, Prout M, Geller AC. Smoking Sleuths: a pilot tobacco prevention elective for medical school students. J Cancer Educ. 2008;23(2):122-5. doi: 10.1080/08858190802039128. PMID 18569248
- [Background] Geller AC, Zapka J, Brooks KR, Dube C, Powers CA, Rigotti N, O'Donnell J, Ockene J; Prevention and Cessation Education Consortium. Tobacco control competencies for US medical students. Am J Public Health. 2005 Jun;95(6):950-5. doi: 10.2105/AJPH.2004.057331. PMID 15914815
- [Background] Linder JA, Rigotti NA, Schneider LI, Kelley JH, Brawarsky P, Haas JS. An electronic health record-based intervention to improve tobacco treatment in primary care: a cluster-randomized controlled trial. Arch Intern Med. 2009 Apr 27;169(8):781-7. doi: 10.1001/archinternmed.2009.53. PMID 19398690
- [Background] Emmons KM, Butterfield RM, Puleo E, Park ER, Mertens A, Gritz ER, Lahti M, Li FP. Smoking among participants in the childhood cancer survivors cohort: the Partnership for Health Study. J Clin Oncol. 2003 Jan 15;21(2):189-96. doi: 10.1200/JCO.2003.06.130. PMID 12525509
- [Background] Park ER, Quinn VP, Chang Y, Regan S, Loudin B, Cummins S, Perry K, Rigotti NA. Recruiting pregnant smokers into a clinical trial: using a network-model managed care organization versus community-based practices. Prev Med. 2007 Mar;44(3):223-9. doi: 10.1016/j.ypmed.2006.10.008. Epub 2007 Jan 3. PMID 17204318
- [Background] Park ER, Puleo E, Butterfield RM, Zorn M, Mertens AC, Gritz ER, Li FP, Emmons KM. A process evaluation of a telephone-based peer-delivered smoking cessation intervention for adult survivors of childhood cancer: the partnership for health study. Prev Med. 2006 Jun;42(6):435-42. doi: 10.1016/j.ypmed.2006.03.004. Epub 2006 Apr 19. PMID 16626797
- [Background] Rigotti NA, Park ER, Regan S, Chang Y, Perry K, Loudin B, Quinn V. Efficacy of telephone counseling for pregnant smokers: a randomized controlled trial. Obstet Gynecol. 2006 Jul;108(1):83-92. doi: 10.1097/01.AOG.0000218100.05601.f8. PMID 16816060
- [Background] Krieger N, Chen JT, Waterman PD, Soobader MJ, Subramanian SV, Carson R. Choosing area based socioeconomic measures to monitor social inequalities in low birth weight and childhood lead poisoning: The Public Health Disparities Geocoding Project (US). J Epidemiol Community Health. 2003 Mar;57(3):186-99. doi: 10.1136/jech.57.3.186. PMID 12594195
- [Background] Ossip DJ, Abrams SM, Mahoney MC, Sall D, Cummings KM. Adverse effects with use of nicotine replacement therapy among quitline clients. Nicotine Tob Res. 2009 Apr;11(4):408-17. doi: 10.1093/ntr/ntp005. Epub 2009 Mar 26. PMID 19325134
- [Background] Baezconde-Garbanati L, Beebe LA, Perez-Stable EJ. Building capacity to address tobacco-related disparities among American Indian and Hispanic/Latino communities: conceptual and systemic considerations. Addiction. 2007 Oct;102 Suppl 2:112-22. doi: 10.1111/j.1360-0443.2007.01962.x. PMID 17850621
- [Background] Luborsky MR. The identification and analysis of themes and patterns. In: Gubrium JF, Sankar A, eds. Qualitative methods in aging research. Thousand Oaks: Sage; 1994.
- [Background] Bernard HR. Social Research Methods: Qualitative and Quantitative Approaches. Thousand Oaks: Sage; 2000.
- [Background] Caraballo RS, Yee SL, Gfroerer JC, Pechacek TF, Henson R. Tobacco use among racial and ethnic population subgroups of adolescents in the United States. Prev Chronic Dis. 2006 Apr;3(2):A39. Epub 2006 Mar 15. PMID 16539780
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2007. MMWR Morb Mortal Wkly Rep. 2008 Nov 14;57(45):1221-6. PMID 19008790
- [Background] Fiore MC, Jaen CR, Baker TB, al. e. Treating Tobacco Use and Dependence: 2008 Update. Rockville, MD: : US Department of Health and Human Services. Public Health Service; 2008.
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Haas JS, Linder JA, Park ER, Gonzalez I, Rigotti NA, Klinger EV, Kontos EZ, Zaslavsky AM, Brawarsky P, Marinacci LX, St Hubert S, Fleegler EW, Williams DR. Proactive tobacco cessation outreach to smokers of low socioeconomic status: a randomized clinical trial. JAMA Intern Med. 2015 Feb;175(2):218-26. doi: 10.1001/jamainternmed.2014.6674. PMID 25506771